CLINICAL TRIAL: NCT00134147
Title: A One Year, Open-Label Outpatient, Parallel Group Trial Assessing the Impact of the Availability of Inhaled Insulin (Exubera) on Glycemic Control in Patients With Type 2 Diabetes Mellitus Who Are Poorly Controlled on a Minimum of Two Oral Anti Diabetic Agents
Brief Title: A Clinical Trial Assessing the Impact of the Availability of Inhaled Insulin on Glucose Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171018
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: Inhaled Insulin

SUMMARY:
To assess the impact on glucose control by inhaled insulin in patients with type 2 diabetes who are not well controlled on 2 or more oral anti-diabetic agents

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 2
* Failing two or more oral anti-diabetic agents

Exclusion Criteria:

* Asthma, COPD
* Smoking

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2005-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin

SECONDARY OUTCOMES:
Percent of patients achieving good control of fasting glucose and lipids
Rate of hypoglycemia
Changes in body weight
Patient satisfaction
Safety based on adverse events reported and laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (111):
- United States (15):
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, San Antonio, Texas
- Canada (10):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Smith Falls, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- France (9):
  - Pfizer Investigational Site, Béthune
  - Pfizer Investigational Site, Bourg-en-Bresse
  - Pfizer Investigational Site, Bron
  - Pfizer Investigational Site, Corbeil-Essonnes
  - Pfizer Investigational Site, La Rochelle
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Roubaix
  - Pfizer Investigational Site, Tours
- Germany (31):
  - Pfizer Investigational Site, Altenburg
  - Pfizer Investigational Site, Aschaffenburg
  - Pfizer Investigational Site, Bad Mergentheim
  - Pfizer Investigational Site, Bad Oeynhausen/ Volmerdingen
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Delmenhorst
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Ebersdorf
  - Pfizer Investigational Site, Eisenach
  - Pfizer Investigational Site, Falkensee
  - Pfizer Investigational Site, Furth im Wald
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Haßloch
  - Pfizer Investigational Site, Künzing
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Meissen
  - Pfizer Investigational Site, Mittweida
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Offenbach
  - Pfizer Investigational Site, Offenburg
  - Pfizer Investigational Site, Oschatz
  - Pfizer Investigational Site, Pirna
  - Pfizer Investigational Site, Riedlhuette
  - Pfizer Investigational Site, Riesa
  - Pfizer Investigational Site, Rossach
  - Pfizer Investigational Site, Schwabenheim
  - Pfizer Investigational Site, St.Ingbert
  - Pfizer Investigational Site, Surwold
  - Pfizer Investigational Site, Wangen
  - Pfizer Investigational Site, Wangen / Allgaeu
  - Pfizer Investigational Site, Witten
- Italy (14):
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Pescara
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Udine
  - Pfizer Investigational Site, Verona
- Spain (11):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, BARCELONA
  - Pfizer Investigational Site, Cadiz, CADIZ
  - Pfizer Investigational Site, Girona, GERONA
  - Pfizer Investigational Site, Granada, GRANADA
  - Pfizer Investigational Site, Las Palmas, LAS Palmas de GRAN Canaria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, SEVILLA
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Barakaldo, VIZCAYA
  - Pfizer Investigational Site, Bilbao, VIZCAYA
- United Kingdom (21):
  - Pfizer Investigational Site, Ayr, Ayrshire
  - Pfizer Investigational Site, Thornhill, Cardiff
  - Pfizer Investigational Site, Penzance, CORNWALL
  - Pfizer Investigational Site, St Austell, Cornwall
  - Pfizer Investigational Site, Truro, Cornwall
  - Pfizer Investigational Site, Plymouth, DEVON
  - Pfizer Investigational Site, Letchworth Garden City, Hertfordshire
  - Pfizer Investigational Site, Sidcup, Kent
  - Pfizer Investigational Site, Whitstable, Kent
  - Pfizer Investigational Site, Blackpool, Lancashire
  - Pfizer Investigational Site, Colney, Norwich
  - Pfizer Investigational Site, Headington, Oxford
  - Pfizer Investigational Site, Penarth, South Glamorgan
  - Pfizer Investigational Site, Dundee, Tayside
  - Pfizer Investigational Site, Haywards Heath, West Sussex
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Bolton
  - Pfizer Investigational Site, Canterbury
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Salford
  - Pfizer Investigational Site, York

REFERENCES:
- [Derived] Freemantle N, Strack TR; Real World Trialists. Will availability of inhaled human insulin (Exubera) improve management of type 2 diabetes? The design of the Real World trial. Trials. 2006 Aug 10;7:25. doi: 10.1186/1745-6215-7-25. PMID 16901335
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171018&StudyName=A%20Clinical%20Trial%20Assessing%20the%20Impact%20of%20the%20Availability%20of%20Inhaled%20Insulin%20on%20Glucose%20Control